CLINICAL TRIAL: NCT06638879
Title: Prospective Study of Tacrolimus Toothpaste for Management of Oral Chronic Graft vs. Host Disease (cGVHD) in Stem Cell Transplant Patients
Brief Title: Tacrolimus Toothpaste for Management of Oral Chronic Graft vs. Host Disease (cGVHD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0687
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Chronic Graft Versus Host Disease Oral
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Topical Tacrolimus Treatment (Experimental)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Participants will receive a tacrolimus treatment via toothpaste application twice daily for three months.

SUMMARY:
This study aims to investigate the use of a novel formulation of tacrolimus, as a toothpaste, in a population of patients with oral chronic graft vs. host disease (cGVHD) as an adjunctive therapy in addition to standard-of-care systemic therapy.

The investigators plan to summarize our findings to add to the current body of literature regarding managing cGVHD, specifically those with oral involvement. Additionally, establishing effective topical application of tacrolimus in the oral cavity will allow for future prospective studies comparing outcomes for these patients with a more traditional standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with oral chronic graft vs. host disease (cGVHD)
* Stable immune suppression within two weeks of enrollment
* Ages > 1 year and < 40 years

Exclusion Criteria:

* Clinically confirmed or suspected herpes simplex virus (HSV) stomatitis
* A recent (within 2 weeks of enrollment) escalation in immune suppression or change in systemic immune suppression of ongoing chronic graft vs. host disease (cGVHD)

Ages: 1 Year to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
The presence of mucosal ulcerations | Three months
  Utilizing the Mucosal Ulceration Index, the patient will be evaluated for the presence of mucosal ulcerations.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Bartlett, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States